CLINICAL TRIAL: NCT03746197
Title: Interactive Digital Technology (Project EVO) to Assess and Improve Cognitive Dysfunction in Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: Interactive Digital Technology to Assess and Improve Cognitive Dysfunction in Patients With Systemic Lupus Erythematosus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Jewish Health (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Akili Interactive Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HS 3063
Record Dates: First submitted 2018-11-01; First posted 2018-11-19 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Lupus; SLE; Cognition; Cognitive Assessment; Videogames
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Project EVO Multi- Treatment (Experimental): Treatment group receives video game device treatment. Participant plays the game for 30 minutes a day, at least five days a week for four weeks.
  Interventions: Device: Project EVO Multi- Treatment
- Control (No Intervention): No contact control

INTERVENTIONS:
Device: Project EVO Multi- Treatment — The EVO platform assesses perceptual discrimination while single-and multi-tasking. Visuomotor tracking involves navigating a character through a dynamically moving environment while avoiding obstacles. EVO uses adaptive algorithms to change game difficulty on a trial by trial and patient by patient basis for the tracking task and discrimination task with real-time feedback.
  Arms: Project EVO Multi- Treatment

SUMMARY:
The purpose of this study is to evaluate whether a short interactive video game device is associated with performance on standard measures of attention and problem solving in patients with systemic lupus erythematosus(SLE). The study is also designed to see if playing the video game for four weeks improves attention and problem solving in patients with SLE.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SLE

Exclusion Criteria:

* Major neurological problems (head trauma, degenerative vascular or metabolic disorder; neoplasm or toxic exposure) prior to SLE
* Major psychiatric disorder prior to SLE
* Major substance abuse
* Pregnant
* Major motor impairment
* High SLE disease activity
* History of learning disability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in mean response time on EVO Monitor | 30 Days
  Average response time (ms) to in game stimuli
Change in response time variability on EVO Monitor | 30 Days
  Compares response time (ms) while single and multi- tasking in EVO game play
Change in EVO performance threshold | 30 days
  Calculation of performance when participant is single vs. multi-tasking
Change in Digit Vigilance Test Scores | 30 Days
  This task measures attention. Scores are based on number of targets found and time to completion. Scores are converted to a t-score based on demographically corrected normative data.
Change in Trail Making Test Scores | 30 days
  This is a test of visual attention and task switching. Scores are based on time to completion and number of errors made. Scores are converted to a t-score based on demographically corrected normative data.
Change in Stroop Test Scores | 30 days
  This examines cognitive flexibility. The participant reads color words or names ink colors from different pages as quickly as possible within a time limit. The test yields three scores based on the number of items completed on each of the three stimulus sheets as well as in interference score. Scores are converted to a t-statistic based on demographically corrected normative data.
Change in Digit Symbol Substitution Scores | 30 days
  The participant scans a key and draws the correct symbol below a the corresponding number. Number of symbols drawn in 120 seconds is converted to a t-statistic using demographically corrected normative data.

CONTACTS AND LOCATIONS:
Locations (1):
- Natinal Jewish Health, Denver, Colorado, United States